CLINICAL TRIAL: NCT04493177
Title: Effect of an Educational Intervention for the Prevention and Management of Overweight and Obesity During the First 18 Months of Life Children and Mothers With Gestational Diabetes in Insured of the Instituto Mexicano Del Seguro Social.
Brief Title: Educational Intervention in the First 18 Months of Life to Prevent/Manage Obesity of Children After Gestational Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Collaborators: Fundacion Rio Arronte (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Rita A. Gomez Diaz, Principal Investigator, Instituto Mexicano del Seguro Social
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R2018-785-079
Record Dates: First submitted 2020-07-17; First posted 2020-07-30 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Gestational Diabetes; Overweight and Obesity
MeSH Terms: conditions — Diabetes, Gestational; Overweight; Obesity | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gestational diabetes intervention (Experimental): All mothers with gestational diabetes will receive 18 months of educational intervention post-partum. They and their offspring will be evaluated at months 1,2,3,6,9,12,15,and 18.
  Interventions: Behavioral: Educational intervention; Other: Conventional treatment Guia de Practica Clinica IMSS-029-08
- No diabetes intervention (Experimental): Mothers without gestational diabetes will receive 18 months of educational intervention post-partum. They and their offspring will be evaluated at months 1,2,3,6,9,12,15,and 18.
  Interventions: Behavioral: Educational intervention; Other: Conventional treatment Guia de Practica Clinica IMSS-029-08
- No diabetes no intervention (Active Comparator): Mothers without gestational diabetes will receive the conventional care for 18 months post-partum. They and their offspring will be evaluated at months 1,2,3,6,9,12,15,and 18.
  Interventions: Other: Conventional treatment Guia de Practica Clinica IMSS-029-08

INTERVENTIONS:
Behavioral: Educational intervention — Monthly 45-minute sessions will be held, including dietary, and physical activity modification, early stimulation, exclusive breastfeeding for 6 months and the proper introduction of foods, and other support for the mother. The sessions will be supported by personalized contact by WhatsApp and programmed telephone calls, in addition to conventional treatment.
  Arms: Gestational diabetes intervention; No diabetes intervention
Other: Conventional treatment Guia de Practica Clinica IMSS-029-08 — Conventional treatment includes some early stimulation, monthly visits for height/weight measurement of the offspring.

SUMMARY:
In order to evaluate the effect of an educational intervention on mothers with gestational diabetes and their offspring in the first 18 months of life, The intervention will be applied to mothers with gestational diabetes, and a group of mothers without diabetes, against a control group with the normal post-partum treatment. Effects on overweight and obesity will be evaluated in both mothers and offspring.

DETAILED DESCRIPTION:
Effect of an education intervention for the prevention and management of overweight and obesity during the first 18 months of life of offspring and mother with gestational diabetes among insured of the Instituto Mexicano del Seguro Social.

ABSTRACT BACKGROUND: According to ENSANUT 2012, 9.7% of children <5 years already are overweight or obese. Recently, an increase was reported in the frequency of overweight and obesity worldwide, beginning at earlier ages, especially in Mexico. The predisposition to chronic diseases in adults may be programmed in the womb ("fetal programming"). Also, women that suffer diabetes during pregnancy have a very high risk (6.4 times more) of developing diabetes in a middle range. The challenge for health personnel dedicated to the care of mother-child pairs is to achieve glycemic control from conception and to identify all the maternal-fetal secondary complications. To carry out compliance with adherence to medical management and/or healthy eating habits would allow us to reduce future overweight, obesity and the incidence of type 2 diabetes in mother-child pairs. Approaching the mother-child pair is a great opportunity to study the intervention, which would allow us not only have a new, useful awareness in the evaluation of educational strategies, but also to apply good practices of healthy habits for the prevention of obesity and to avoid progression to diabetes. For the aforementioned reasons, the objective is: to implement and evaluate the effect of an education intervention for the prevention and management of overweight and obesity during the first 18 months of life of child and in mothers with and without gestational diabetes in insured members of the Instituto Mexicano del Seguro Social.

MATERIAL AND METHODS. Pregnant women will be invited to participate, who receive their prenatal and/or birth care in the Unidad Médica de Alta Especialidad (UMAE) Gineco-Obstretric Hospital No. 4 (HGO #4) and UMAE HGO #3 of Centro Médico "La Raza" of IMSS. After acceptance and signing an informed consent to participate in the study, 645 mother-child pairs will be included, with and without gestational diabetes mellitus (GDM), which will be diagnosed according to the criteria of the American Diabetes Association; all mothers with be between 18 and 40 years old. There will be 3 groups of binomials: 1) with GDM, 2) without GDM who will received the education intervention, and 3) without GDM who will receive the conventional care IMSS offers to mothers and nursing infants, during the first 18 months post-partum.

At the time of canalization before delivery or cesarean, a blood sample (15 mL) will be taken from the mother for measurement of glucose, glucosylated hemoglobin (A1c) and lipid profile. After birth, blood (15 mL) will be extracted directly from the umbilical cord for measurement of the child's glucose and lipid profile. Once the pediatric doctor has carried out reanimation of the newborn, previously-standardized health staff will take anthropometric measurements. During the 18 months of follow-up from birth, the mother-child pair will be given appointments at 0, 1, 2, 3, 6, 9, 12, 15 and 18 months, in which health care personnel involved in the study (nutritionist, social worker, pediatrician and family doctor) will perform activities to promote health and prevent disease, directed towards the mother-child pair and planned within the education intervention strategy based on the First 1000 Days program, or the conventional care that mothers and nursing infants receive in IMSS, according to the study group. Weekly, the mothers will be sent, by digital media and social networks, educational material to promote healthy diet and physical activity; for the child material will include the promotion of exclusive breastfeeding until 6 months, at which time promotion will be of adequate complementary foods, in addition to early stimulation activities; educational material will be handed out: posters and brochures will serve to reinforce and remind of the information given during appointments. Also, characteristics of the diet consumed by mother and child will be recorded monthly, along with the physical activity performed by the mother.

The education intervention has as objective the acquiring of knowledge, motivation, creation of an awareness of disease, adoption of healthy diet and physical activity; its components will be individual sessions, group sessions, electronic messages, etc.

SAMPLE SIZE: The sample size necessary, with a 95% confidence interval and a power of 80%, is 645 mother-child pairs, among which 215 mother-child pairs will be included with mothers who presented gestational diabetes and will receive the education intervention, and 430 pairs without gestational diabetes (215 pairs with the education intervention and 215 with conventional care).

STATISTICAL ANALYSIS: Anthropometric and biochemical data will be described using mean and standard deviation for continuous variables, or percentages for nominal or ordinal variables. The difference between variables of offspring of mothers with and without GDM, as well as the difference between groups with and without education intervention, will be analyzed with Mann-Whitney U test, Student t test, or chi square, as appropriate. Multivariate analysis will be performed, using lineal regression in models of repeated measures, to evaluate the association between 1) child weight-for-age (in Z score), and 2) mother's BMI, and the education intervention or having presented GDM or no, according to the independent variable, or the exposure that is being analyzed (effect of GDM or effect of the intervention), controlling for possible confounding variables. Values of p<0.05 will be considered statistically significant.

EXPECTED RESULTS: The education intervention was standardized in Boston, Mass, and will be implemented with the adaptation necessary for our population, in order to evaluate if it is better than the conventional treatment, for transference to the Family Medicine Units and second-level hospitals that have Gineco-obstetric services in the IMSS.

Included will be surveys on the opinion of doctors and participants to measure the acceptability of the intervention.

Expected results are: differences associated with the intervention in: a) body mass index and weight-for-age, respectively, in the mother-child pair; b) speed of growth and growth percentile score; as well as c) implementation of an education strategy that can be used as part of the care the mother-child pair receives.

DELIVERABLE PRODUCTS: Situational analysis of the mother-child pair, from the clinical point of view, laboratory studies, databases, plan for implementation of this strategy in IMSS. In addition, there will be databases that can be used for other analyses. DNA banks are contemplated, from serum and plasma, for scientific questions derived from this study.

SOCIAL IMPACT: This study will offer a model that can be implemented in all hospitals of IMSS that attend to births and/or cesareans. This will contribute to the timely prevention of obesity in insured families of IMSS, with an eye towards making it extend both at the national level for IMSS and for other health institutions. It is hoped that the education strategy will be a tool that allows a reduction in the frequency of overweight, obesity, and diabetes mellitus in our country.

DURATION OF THE STUDY: 2 years.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* insured by IMSS
* with or without gestational diabetes

Exclusion Criteria:

* History of type 1 or 2 diabetes, MODY or secondary diabetes
* CKD, hepatic or cardiac disease, pregnancy hypertension, corioamniotis orpremature membrane rupture, pulmonary maturity 24 hours before birth, severe complications

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 645 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-08-25 (Estimated)

PRIMARY OUTCOMES:
Prevention of overweight/obesity in offspring, determined by z-score in the indicator for weight for age | 18 months
  Offspring will be expected to have a difference of at least 0,3 standard deviations in z-score of the indicator for weight for age, as measured by weight on a standard weight scale over the course of the study, and compared with WHO growth charts.
Prevention of overweight/obesity mothers, determined by loss in body mass index (BMI) | 18 months
  Mothers will be expected to have a loss of at least 1.8kg/m2 of body mass index (BMI, weight/height squared), as measured by weight, as measured by a standard weight scale, divided by height in meters squared over the course of the study.

SECONDARY OUTCOMES:
Changes in blood concentration of glucose: GDM | 18 months
  Compare blood measurements of glucose of the mother over the 18 months of mothers with vs without gestational diabetes (GDM).
Changes in blood concentration of glucose: intervention | 18 months
  Compare blood measurements of glucose of the mother over the 18 months of mothers with vs without educational intervention.
  .
Changes in blood concentration of glycosylated hemoglobin: GDM | 18 months
  Compare blood measurements of glycosylated hemoglobin (HbA1c) of the mother over the 18 months of mothers with vs without gestational diabetes.
  .
Changes in blood concentration of glycosylated hemoglobin: intervention | 18 months
  Compare blood measurements of glycosylated hemoglobin (HbA1c) of the mother over the 18 months of mothers with vs without educational intervention.
  .
Changes in blood concentration of lipids: GDM | 18 months
  Compare blood measurements of lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides) of the mother over the 18 months of mothers with vs without gestational diabetes.
  .
Changes in blood concentration of lipids: intervention | 18 months
  Compare blood measurements of lipid profile (total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides) of the mother over the 18 months of mothers with vs without educational intervention.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Cesar R Gonzalez Bonilla, PhD, Study Chair — Secretary of Health
Locations (1):
- Hospital Gineco-Obstetrico #4, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Research will be shared upon written request.

REFERENCES:
- [Derived] Soto Briseno AI, Gomez-Diaz RA, Saldana Espinoza RC, Lavielle P, Valdez Gonzalez AL, Wacher NH. Validation of the COVID-19 Fear Scale modified for application during the perinatal period. J Psychosom Obstet Gynaecol. 2022 Dec;43(4):447-452. doi: 10.1080/0167482X.2022.2050210. Epub 2022 Mar 16. PMID 35294335